CLINICAL TRIAL: NCT00468364
Title: Comparison of Carbohydrate Metabolism During the Night and at Hypoglycemia in Type-2 Diabetic Patients Either on Glargine or NPH Insulin
Brief Title: Comparison of Insulin Glargine and NPH Insulin at Night and at Hypoglycemia in Type 2 Diabetes
Acronym: ClampHOE901
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Collaborators: Sanofi (Industry)
Other Study IDs: Clamp EC 48/2003
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Last update posted 2007-08-30 (Estimated); Status verified 2007-08

CONDITIONS: Diabetes
Keywords: Hypoglycemia, bedtime insulin, long-acting insulin
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia | interventions — Insulin Glargine; Insulin, Isophane

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin glargine
Drug: NPH insulin

SUMMARY:
Long-acting insulin injected at bedtime may cause hypoglycemia (low blood sugar) in the night in patients with diabetes. The aims of the study are 1) to compare the dynamic characteristics of long-acting insulin analog glargine with those of NPH insulin and placebo during the night and the early morning hours, 2) investigate differences on glucose metabolism of bedtime glargine versus NPH insulin at induced hypoglycemia.

DETAILED DESCRIPTION:
Patients with advanced type 2 diabetes like those with type 1 diabetes are at risk for defective glucose counterregulation and hypoglycemia unawareness, the components of hypoglycemia-associated autonomic failure and the resultant vicious cycle of recurrent iatrogenic hypoglycemia. This may explain why iatrogenic hypoglycemia becomes limiting to glycemic control as patients approach the insulin-deficient end of the spectrum of type 2 diabetes. Compared to Neutral Protamin Hagedorn (NPH) insulin glargine is a new long-acting peakless analogue with lower incidence of nocturnal hypoglycemia having the potential to decrease the frequency of hypoglycemia of insulin therapy. Modern type 2 diabetes therapy guidelines recommend insulin for an increasing population of patients. There is no doubt that type 2 diabetic patients suffer from hypoglycemia under insulin therapy, however it is not clear whether the extensive studies on hypoglycemia in type 1 patients apply also for type 2 diabetes. Recent reports indicate that type 2 diabetic patients of long duration react similarly to a hypoglycemic clamp as type 1 diabetic patients while well controlled type 2 diabetics had even more favorable thresholds for counter-regulatory hormone secretion. On the basis of these considerations the aims of this study are to 1) more precisely define the mechanisms of hypoglycemia in type 2 diabetes, 2) to investigate differences on glucose and lactate metabolism of bedtime NPH insulin versus glargine. To address these objectives we will use the hypoglycemic clamping technique combined with infusion of stable isotopes of glucose and lactate and non-invasive measurement of muscle flow characteristics at hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes mellitus
* Therapy may be with either insulin alone or in combination with oral anti-diabetic agents
* Metabolic control with HbA1c values < 10%

Exclusion Criteria:

* Other than type 2 diabetes
* Pregnancy
* Systemic Corticosteroids, Beta-blockers
* Clinically relevant cardiovascular, gastrointestinal, hepatic, neurologic, endocrine, haematological or other major disease making implementation of the protocol or interpretation of the study results difficult
* History of drug or alcohol abuse
* Impaired renal function (serum creatinine > 1.3 mg/dl)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-07; Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Linn, MD, Principal Investigator — Justus Liebig University
Locations (1):
- Clinical Research Unit, Giessen, Germany

REFERENCES:
- [Background] Yki-Jarvinen H, Kauppinen-Makelin R, Tiikkainen M, Vahatalo M, Virtamo H, Nikkila K, Tulokas T, Hulme S, Hardy K, McNulty S, Hanninen J, Levanen H, Lahdenpera S, Lehtonen R, Ryysy L. Insulin glargine or NPH combined with metformin in type 2 diabetes: the LANMET study. Diabetologia. 2006 Mar;49(3):442-51. doi: 10.1007/s00125-005-0132-0. Epub 2006 Feb 3. PMID 16456680